CLINICAL TRIAL: NCT04347213
Title: The Link Between Omnivorous, Vegan, Vegetarian, Low Carb Diets and Health Indicators in Healthy Subjects With Normal Weight
Brief Title: The Link Between Diets and Health Indicators
Acronym: DIETE
Status: Completed | Type: Observational
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, associate professor, University of Primorska
Other Study IDs: DIETE
Record Dates: First submitted 2020-04-03; First posted 2020-04-15 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Healthy Diet; Microbiota
Keywords: diet; gut microbiota; longevity; inflammation; health
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole blood and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- omnivors: Participants who habitually consume all food groups in their diet.
  Interventions: Behavioral: Regular lifestyle in different circumstances
- vegetarian: Participants who habitually avoid meat in their diet.
  Interventions: Behavioral: Regular lifestyle in different circumstances
- vegan: Participants who habitually avoid all animal source food in their diet.
  Interventions: Behavioral: Regular lifestyle in different circumstances
- low-carbohydrate high-fat diet: Participants who habitually avoid carbohydrate in their diet.
  Interventions: Behavioral: Regular lifestyle in different circumstances

INTERVENTIONS:
Behavioral: Regular lifestyle in different circumstances — Participants' lifestyle will be followed over the years.

SUMMARY:
The cohort study investigates the effect of different dietary intake among omnivorous, vegan, vegetarian and low-carb diets on health parameters and on long-term overall health. The participants blood parameters, dietary intake, gut microbiota composition, body mass and composition, resting energy expenditure, lifestyle factors and psychological factors will be determined and measured.

DETAILED DESCRIPTION:
Vegetarian and vegan diets have been shown to have health benefits on preventing cardiovascular diseases, type 2 diabetes and cancer. They are both gaining popularity in public. Ketogenic diet has also been very popular, especially due to its effect on weight loss and blood glucose parameters. To our knowledge there, are no studies that compare long-term effects of all three diets and omnivorous diets with regards to health parameters and gut microbiota composition.

The aim of the proposed study is to investigate the link between different diets and health parameters, such as parameters related to longevity, inflammation, stress and gut microbiota composition. The study is designed to compare different diets and their relationship with the body as a whole.

ELIGIBILITY:
Inclusion Criteria:

* 18,5 < BMI < 30 kg/m2
* asymptomatic for any disease
* medication free
* same pattern of eating in the last 3 months
* stable body mass in the last 3 months

Exclusion Criteria:

* BMI < 18,5 and > 30 kg/m2
* presence of any chronic disease
* taking any medications
* changed eating pattern in the last 3 months
* unstable body mass in the last 3 months
* taking antibiotics in the last 3 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals with stable body mass with specific eating patterns: omnivores, vegetarians, vegan, low carb high fat.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Changes in systemic inflammation | Change from baseline at 5 years.
  CRP [mg/L] will be measured as a marker of inflammation.
Changes in serum total antioxidative capacity | Change from baseline at 5 years.
  Total antioxidative capacity of serum will be measured with Photochem instrument and expressed as nanomole equivalents of ascorbic acid per microliter of serum.

SECONDARY OUTCOMES:
Changes in macronutrient intake | Change from baseline at 5 years.
  Macronutrient intake will be measured with validated FFQ and 3-day food diary and analysed with softwares OPEN and Prodi. Macronutrient intake will be expressed as part of daily energy intake.
Changes in micronutrient intake | Change from baseline at 5 years.
  Micronutrient intake will be measured with validated FFQ and 3-day food diary and analysed with softwares OPEN and Prodi. Micronutrient intake will be expressed as mg per day.
Changes in gut microbiota composition | Change from baseline at 5 years.
  Microbial composition of stool will be determined with microbial DNA isolation and identification.
Changes in body composition | Change from baseline at 5 years.
  Fat free body mass will be measured with bioelectrical impedance analysis and expressed in kg.
Changes in resting metabolic rate | Change from baseline at 5 years.
  Resting metabolic rate will be determined with indirect calorimeter and expressed in kJ/day.
Changes in lifestyle factors | Change from baseline at 5 years.
  Will be assessed with a questionnaire.
Changes in anxiety | Change from baseline at 5 years.
  Will be assessed by state-trait anxiety inventory. The STAIX-1 contains 20 items, which are scored on a 4-pointscale with subscale scores ranging from 20 to 80, with higherscores indicating higher anxiety.
Changes in body satisfaction | Change from baseline at 5 years.
  Will be assessed by the body dissatisfaction subscale from the Eating Disorders Inventory-2. Responses will be rated on a 5-point Likert scale from 0 (never) to 4 (always).
Changes in grip strength | Change from baseline at 5 years.
  Will be measured with a hand dynamometer.
Changes in autophagy | Change from baseline at 5 years.
  Autophagy will be measured by autophagy-related mRNA gene expression evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Zala Jenko Pražnikar, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences; Nina Mohorko, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paoli A, Mancin L, Bianco A, Thomas E, Mota JF, Piccini F. Ketogenic Diet and Microbiota: Friends or Enemies? Genes (Basel). 2019 Jul 15;10(7):534. doi: 10.3390/genes10070534. PMID 31311141
- [Background] Rocha JP, Laster J, Parag B, Shah NU. Multiple Health Benefits and Minimal Risks Associated with Vegetarian Diets. Curr Nutr Rep. 2019 Dec;8(4):374-381. doi: 10.1007/s13668-019-00298-w. PMID 31705483
- [Background] Sakkas H, Bozidis P, Touzios C, Kolios D, Athanasiou G, Athanasopoulou E, Gerou I, Gartzonika C. Nutritional Status and the Influence of the Vegan Diet on the Gut Microbiota and Human Health. Medicina (Kaunas). 2020 Feb 22;56(2):88. doi: 10.3390/medicina56020088. PMID 32098430
- [Background] Satija A, Bhupathiraju SN, Rimm EB, Spiegelman D, Chiuve SE, Borgi L, Willett WC, Manson JE, Sun Q, Hu FB. Plant-Based Dietary Patterns and Incidence of Type 2 Diabetes in US Men and Women: Results from Three Prospective Cohort Studies. PLoS Med. 2016 Jun 14;13(6):e1002039. doi: 10.1371/journal.pmed.1002039. eCollection 2016 Jun. PMID 27299701
- [Background] Kenig S, Petelin A, Poklar Vatovec T, Mohorko N, Jenko-Praznikar Z. Assessment of micronutrients in a 12-wk ketogenic diet in obese adults. Nutrition. 2019 Nov-Dec;67-68:110522. doi: 10.1016/j.nut.2019.06.003. Epub 2019 Jun 14. PMID 31445313
- [Background] Mohorko N, Petelin A, Jurdana M, Biolo G, Jenko-Praznikar Z. Elevated serum levels of cysteine and tyrosine: early biomarkers in asymptomatic adults at increased risk of developing metabolic syndrome. Biomed Res Int. 2015;2015:418681. doi: 10.1155/2015/418681. Epub 2015 Mar 4. PMID 25821801
- [Background] Mohorko N, Jenko-Praznika Z, Petelin A. Leucine and lysine intakes are highly associated with serum adiponectin levels in asymptomatic adults. Minerva Endocrinol. 2016 Sep;41(3):302-13. Epub 2015 Feb 13. PMID 25677829
- [Background] Cernelic-Bizjak M, Jenko-Praznikar Z. Body dissatisfaction predicts inflammatory status in asymptomatic healthy individuals. J Health Psychol. 2018 Jan;23(1):25-35. doi: 10.1177/1359105316672923. Epub 2016 Oct 19. PMID 28810361
- [Background] Bizjak M, Jenko-Praznikar Z, Korousic Seljak B. Development and validation of an electronic FFQ to assess food intake in the Slovene population. Public Health Nutr. 2014 Aug;17(8):1729-37. doi: 10.1017/S1368980013002577. Epub 2013 Oct 8. PMID 24103359
- [Background] Jenko-Praznikar Z, Petelin A, Jurdana M, Ziberna L. Serum bilirubin levels are lower in overweight asymptomatic middle-aged adults: an early indicator of metabolic syndrome? Metabolism. 2013 Jul;62(7):976-85. doi: 10.1016/j.metabol.2013.01.011. Epub 2013 Feb 13. PMID 23414908
- [Derived] Bogataj Jontez N, Kenig S, Sik Novak K, Petelin A, Jenko Praznikar Z, Mohorko N. Habitual low carbohydrate high fat diet compared with omnivorous, vegan, and vegetarian diets. Front Nutr. 2023 Apr 13;10:1106153. doi: 10.3389/fnut.2023.1106153. eCollection 2023. PMID 37125046
- [Derived] Sik Novak K, Bogataj Jontez N, Kenig S, Hladnik M, Baruca Arbeiter A, Bandelj D, Cernelic Bizjak M, Petelin A, Mohorko N, Jenko Praznikar Z. The effect of COVID-19 lockdown on mental health, gut microbiota composition and serum cortisol levels. Stress. 2022 Jan;25(1):246-257. doi: 10.1080/10253890.2022.2082280. PMID 35713539